CLINICAL TRIAL: NCT00691249
Title: Resistant Starch on Glucose and Insulin Sensitivity in Individuals With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kansas State University (Other)
Collaborators: MGP Ingredients, Inc. (Industry)
Responsible Party: Mark Haub Ph.D., Department of Human Nutrition
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: KSU-HML-RSt3
Record Dates: First submitted 2008-05-22; First posted 2008-06-05 (Estimated); Last update posted 2009-07-02 (Estimated); Status verified 2008-05

CONDITIONS: Hyperglycemia
Keywords: Diabetes; Diet; Fiber
MeSH Terms: conditions — Hyperglycemia; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental): Resistant starch type 4-Raw
  Interventions: Dietary Supplement: Resistant Starch Type 4-Raw
- 2 (Experimental): Resistant starch type 4-Raw
  Interventions: Dietary Supplement: Resistant Starch Type 4-Raw
- 3 (Experimental): Resistant starch type 4-Cooked
  Interventions: Dietary Supplement: Resistant Starch Type 4-Cooked
- 4 (Experimental): Resistant starch type 4-Cooked
  Interventions: Dietary Supplement: Resistant Starch Type 4-Cooked
- 5 (Placebo Comparator): Shredded wheat
  Interventions: Dietary Supplement: Shredded Wheat

INTERVENTIONS:
Dietary Supplement: Resistant Starch Type 4-Raw — Low Dose- 70g bar
  Arms: 1
Dietary Supplement: Resistant Starch Type 4-Raw — High Dose- 100g bar
  Arms: 2
Dietary Supplement: Resistant Starch Type 4-Cooked — Low Dose- 70g bar
  Arms: 3
Dietary Supplement: Resistant Starch Type 4-Cooked — High dose: 100g bar
  Arms: 4
Dietary Supplement: Shredded Wheat — 70g bar
  Arms: 5

SUMMARY:
This study will test the effects of resistant starch type 4 on blood sugar and hunger in adults with Type 2 diabetes.

DETAILED DESCRIPTION:
To measure the blood glucose response, after an overnight fast, blood samples will be collected before eating and 15, 30, 45, 60, 90, and 120 minutes after eating each bar. The incremental area under the curve was used to calculate glycemic index. The investigators will also measure the second meal effect by measuring the metabolic response (glucose, insulin, and gut hormones) after a standardized lunch two hours following the first assessment.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetics

Exclusion Criteria:

* Diagnosed with other metabolic disorders
* Allergies to wheat
* Non-smokers

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Post-Prandial metabolism | Acute -- fasting, 15, 30, 45, 60, 90 and 120 minutes post-ingestion

SECONDARY OUTCOMES:
Satiety | Early morning - Midafternoon

CONTACTS AND LOCATIONS:
Overall Officials: Mark Haub, Ph.D., Principal Investigator — Department of Human Nutrition
Locations (1):
- Kansas State Univerity: Department of Human Nutrition, Manhattan, Kansas, United States